CLINICAL TRIAL: NCT03072524
Title: Validation of Prehospital Stroke Scale (FAST PLUS TEST) to Predict Patients With Large Arterial Vessel Intracranial Occlusion.
Brief Title: The Prehospital Selection of Acute Stroke Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); Agel Research and Training Institute (Other); Emergency Medical Service Ostrava, Ostrava, Czech Republic (Unknown); Municipal Hospital Ostrava, Ostrava, Czech Republic (Unknown); St. Anne's University Hospital Brno, Czech Republic (Other); Angels Initiative, European Stroke Organisation, Czech branch (Unknown)
Responsible Party: Sponsor
Other Study IDs: FNO-NK-1
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: pre-hospital stroke scale test; severe hemiparesis; large vessel occlusion; mechanical thrombectomy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Stroke patients who will undergo the FAST PLUS test within 12 hours from the stroke onset.
  Interventions: Diagnostic Test: FAST PLUS test

INTERVENTIONS:
Diagnostic Test: FAST PLUS test — FAST PLUS test consists of two parts: the first one is the standard FAST test, which evaluates Speech (0-1), Facial palsy (0-1), Arm motor function (0-1), Time (0-1). The second part of the FAST PLUS test evaluates only the presence of severe arm or leg motor deficit (0-1), and unilateral occurrence of this motor function deficit (0-1).

SUMMARY:
The aim of this study is to develop and validate a simple prehospital stroke scale, which would predict the presence of large vessel occlusion (LVO) in patients with acute stroke. This study prospectively evaluates the predictive value of a new simple pre-hospital scale (FAST PLUS test) for the presence of large vessel occlusion in anterior intracranial circulation. The FAST PLUS test consists of two parts: the first is the well-known FAST test, which is employed in all possible cases of stroke occurrence. This test consists of the following items: Speech (scored 0-1), Facial palsy (0-1), any failure of Arm motor function (0-1), and Time (0-1). The second part of FAST PLUS test evaluates only the presence of severe arm or leg motor deficit (scored 0-1) and unilateral occurrence of its motor function deficit (scored 0-1).

The FAST PLUS test will be used prospectively at the place of stroke onset by trained medical emergency technicians. The first objective of study is to evaluate the sensitivity, specificity, and the positive and negative predictive value of the test which relate to the presence of occlusion of intracranial artery (intracranial carotid artery, T occlusion and occlusion of Middle Cerebral artery segment M1 and M2). CT angiography can only diagnose the LVO.

The second objective of this study is to assess inter-rater variability among stroke specialists and emergency technicians, concerning the presence of severe motor arm or leg deficit.

The third objective : After implementation of the FAST TEST to clinical practice, we aim to achieve the acceleration of transport time in FAST PLUS positive patients via direct transport to Comprehensive Stroke Center to mechanical thrombectomy.

DETAILED DESCRIPTION:
The effective treatment of acute ischemic stroke is limited to administration of intravenous tissue-type plasminogen activator within the first 4.5 hours from symptoms onset or endovascular thrombectomy up to 6(8) hours from the symptoms onset. Intravenous thrombolysis can be administered in the nearest Primary Stroke Centers (PSC).

In the case of large vessel occlusion, the endovascular therapy (mechanical thrombectomy) is utilized. Mechanical thrombectomy is offered only in Comprehensive Stroke Centers (CSC), due to the necessary presence of the special endovascular team during the procedure.

Practically, there are two options to transport patients for endovascular treatment. If the first one is used, then all suspected stroke patients are transported to primary stroke centers only. Then, rapid examinations are provided and, if the patient is determined to be having a stroke, the administration of intravenous thrombolysis occurs. Patients with diagnosis of stroke and large vessel occlusion are consequently transported to Comprehensive Stroke Center in order to receive mechanical thrombectomy. This first choice accelerates thrombolysis administration but delays endovascular procedures.

The second option entails selection of patients with suspected LVO stroke on site of stroke onset, and such patients are directly transported to Comprehensive Stroke Centers. The second choice accelerates endovascular procedures, but may delay intravenous thrombolysis. The disadvantage of this might be the overloading of the CSC with misdiagnosed patients (stroke mimics or non LVO stroke patients).

We can identify suspected stroke patients pre-hospitably with relative accuracy. The FAST test is a very simple and highly specific tool to identify stroke patients.* It consists of four items Face, Arm, Speech, and Time. Unfortunately, the FAST test is not able to evaluate the severity of the stroke, which is probably linked to the occlusion of large artery.

The only one test (RACE test) was prospectively studied to evaluate its sensitivity and specificity for diagnosis of large vessel occlusion.

In the hospital (stroke centre), we recognize the stroke severity according to NIHS scale, but both these scales are not suitable for emergency service for its difficulty.

Therefore, we desined a very simple new test - FAST PLUS test for the identification of the severe stroke patients on site, immediately at the onset of stroke. FAST PLUS test consists of two parts: the first one is the well-known FAST test which selects all suspected stroke patients and consists of the following evaluations: Speech (scored 0-1), Facial palsy (0-1), any failure of Arm motor function (0-1), time (0-1). The time means the speed of onset of symptoms during 30 minutes. The second part of the FAST PLUS test evaluates only the presence of severe arm or leg motor deficit (scored 0-1) and the unilateral occurrence of this motor function deficit (scored 0-1). (Figure one) The working hypothesis: We assume that the patients with clinically severe stroke and positive FAST PLUS test have a high probability of the presence of large cerebral vessel occlusion.

The aims of study:

A) The validation of the new pre-hospital test - FAST PLUS - to identify the stroke patients with LVO. The objective of our study is to evaluate the predictive value of the FAST PLUS test in the detection of patients with acute stroke and large vessel occlusion (LVO) when it is used by medical emergency technicians during the pre-hospital phase.

We presume that stroke severity, according to item 4 and 5 in NIHSS is linked to occlusion of ACM M1 or intracranial ICA. The FAST PLUS test consists of two parts (fig. 1), the first one is FAST test for identifying patients with stroke. The second part of test has three items, and evaluates the severity of hemiparesis and unilateral disabilities. The FAST PLUS test is positive when at least two items are positive in the first part (Time must be always positive + the presence of one of three symptoms at least) and all three items are positive in the second part.

B) The second aim of study is to determine the inter-rater variability between emergency technician and stroke specialist in evaluation NIHS scale, items 4 and 5 only. The agreement means the agreement in the severe hemiparesis evaluation between paramedics (FAST PLUS test positive) and stroke specialist examination(NIHSS 3 or 4 points in item 4,5 NIHSS) .

C) The third aim of study is to shorten the time between the onset of stroke to hospital entry or the time from the arriving of emergency service on site of stroke to hospital door after implementation of FAST PLUS test to the daily medical practice.

The first phase:

The creation of educational material for emergency technicians. The second phase: The education and testing of emergency technicians via e-learning and web seminars. The aim of the education is to learn whether the Emergency service is using the FAST PLUS test correctly.

We plan 6 months time period for the first and the second phase of study.

The third phase:

A/ to collect 400 FAST PLUS tests from the stroke patients up to 12 hours from the stroke onset to hospital arrival.

B/ to calculate the primary secondary and tertiary outcome measures of study

We plan 12 months time period for the third phase of study.

For statistical analysis, X software was used. Receiver operating curves and areas under receiver operating curve (c-statistics) were calculated as a measure of predictive ability for LVO of the FAST plus test. Ideal prediction produces a c-statistic of 1.00; precision no better than chance is associated with c-statistic of ≤0.50. Correlation between both scales (FAST test second part and NIHSS items 4 and 5) was analyzed with the nonparametric Spearman coefficient.

Cross tables for different cutoff values of the FAST plus test were used to evaluate sensitivity, specificity, positive predictive value, negative predictive values, and overall accuracy for the presence of VO.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* FAST PLUS test evaluation performed by emergency technicians
* CT,CT angiography evaluation performed up to 12 hours from stroke onset

Exclusion Criteria:

* Non ischemic stroke etiology of acute neurological deficit
* More than 12 hours from the symptoms onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-hospital suspected stroke patients according to FAST PLUS test.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive, negative predictive value and accuracy | 21 months
  Sensitivity, specificity, positive, negative predictive value of the test and overall accuracy with the presence of large vessel occlusion will be assessed. The presence of LVO will be diagnosed by CT Angiography only as soon as the patient enters the hospital.

SECONDARY OUTCOMES:
Inter-rater variability | 21 months
  Inter-rater variability between emergency technicians and stroke specialist in stroke severity (hemiparesis) assessment.

OTHER OUTCOMES:
Time to hospital | 21 months
  The time from the arriving of emergency service on site of stroke to door of hospital (comprehensive stroke center) after implementation of FAST PLUS test to the daily medical practice. We compare the time before and after the implementation of FAST PLUS test to daily clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Bar, Ass.Prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (4):
- Czechia (4):
  - Emergency Medical Service Ostrava, Ostrava, Moravian-Silesian Region
  - Ostrava University, Ostrava, Moravian-Silesian Region
  - Agel Research and Training Institute, Ostrava Vitkovice Hospital, Czech Republic, Ostrava, Moravian-Silesian Region
  - Municipal Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez de la Ossa N, Carrera D, Gorchs M, Querol M, Millan M, Gomis M, Dorado L, Lopez-Cancio E, Hernandez-Perez M, Chicharro V, Escalada X, Jimenez X, Davalos A. Design and validation of a prehospital stroke scale to predict large arterial occlusion: the rapid arterial occlusion evaluation scale. Stroke. 2014 Jan;45(1):87-91. doi: 10.1161/STROKEAHA.113.003071. Epub 2013 Nov 26. PMID 24281224
- [Background] Nazliel B, Starkman S, Liebeskind DS, Ovbiagele B, Kim D, Sanossian N, Ali L, Buck B, Villablanca P, Vinuela F, Duckwiler G, Jahan R, Saver JL. A brief prehospital stroke severity scale identifies ischemic stroke patients harboring persisting large arterial occlusions. Stroke. 2008 Aug;39(8):2264-7. doi: 10.1161/STROKEAHA.107.508127. Epub 2008 Jun 12. PMID 18556587
- [Background] Singer OC, Dvorak F, du Mesnil de Rochemont R, Lanfermann H, Sitzer M, Neumann-Haefelin T. A simple 3-item stroke scale: comparison with the National Institutes of Health Stroke Scale and prediction of middle cerebral artery occlusion. Stroke. 2005 Apr;36(4):773-6. doi: 10.1161/01.STR.0000157591.61322.df. Epub 2005 Feb 24. PMID 15731478
- [Background] Puolakka T, Kuisma M, Lankimaki S, Puolakka J, Hallikainen J, Rantanen K, Lindsberg PJ. Cutting the Prehospital On-Scene Time of Stroke Thrombolysis in Helsinki: A Prospective Interventional Study. Stroke. 2016 Dec;47(12):3038-3040. doi: 10.1161/STROKEAHA.116.014531. Epub 2016 Nov 8. PMID 27827326
- [Background] Lima FO, Silva GS, Furie KL, Frankel MR, Lev MH, Camargo EC, Haussen DC, Singhal AB, Koroshetz WJ, Smith WS, Nogueira RG. Field Assessment Stroke Triage for Emergency Destination: A Simple and Accurate Prehospital Scale to Detect Large Vessel Occlusion Strokes. Stroke. 2016 Aug;47(8):1997-2002. doi: 10.1161/STROKEAHA.116.013301. Epub 2016 Jun 30. PMID 27364531
- [Background] Heldner MR, Zubler C, Mattle HP, Schroth G, Weck A, Mono ML, Gralla J, Jung S, El-Koussy M, Ludi R, Yan X, Arnold M, Ozdoba C, Mordasini P, Fischer U. National Institutes of Health stroke scale score and vessel occlusion in 2152 patients with acute ischemic stroke. Stroke. 2013 Apr;44(4):1153-7. doi: 10.1161/STROKEAHA.111.000604. Epub 2013 Mar 7. PMID 23471266
- [Background] Hastrup S, Damgaard D, Johnsen SP, Andersen G. Prehospital Acute Stroke Severity Scale to Predict Large Artery Occlusion: Design and Comparison With Other Scales. Stroke. 2016 Jul;47(7):1772-6. doi: 10.1161/STROKEAHA.115.012482. Epub 2016 Jun 7. PMID 27272487
- [Background] Meyer BC, Lyden PD. The modified National Institutes of Health Stroke Scale: its time has come. Int J Stroke. 2009 Aug;4(4):267-73. doi: 10.1111/j.1747-4949.2009.00294.x. PMID 19689755
- [Background] Harbison J, Hossain O, Jenkinson D, Davis J, Louw SJ, Ford GA. Diagnostic accuracy of stroke referrals from primary care, emergency room physicians, and ambulance staff using the face arm speech test. Stroke. 2003 Jan;34(1):71-6. doi: 10.1161/01.str.0000044170.46643.5e. PMID 12511753
- [Derived] Vaclavik D, Bar M, Klecka L, Holes D, Cabal M, Mikulik R. Prehospital stroke scale (FAST PLUS Test) predicts patients with intracranial large vessel occlusion. Brain Behav. 2018 Sep;8(9):e01087. doi: 10.1002/brb3.1087. Epub 2018 Aug 7. PMID 30085409
- See also: An initiative by national and international government entities, private and scholastic organizations, dedicated to promoting wellness and better patient care in the field of stroke. — http://www.nihstrokescale.org/
- See also: Stroke reports clinical and experimental information on the prevention, diagnosis, and treatment of cerebrovascular diseases. — http://stroke.ahajournals.org